CLINICAL TRIAL: NCT05805020
Title: Is There a Concordance Between the Cellvizio With an Intravenous Injection of Fluorescein and the Pathology to Determine the Microscopic Inflammation at the Ileal Resection Margins in Crohn's Ileal Disease
Brief Title: Cellvizio to Evaluate Margins in Crohn's Ileal Disease
Acronym: CELLVICROHN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2022_843_0111
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Resection Margins; Recurrence
Keywords: Crohn Disease; Resection Margins; recurrence
MeSH Terms: conditions — Crohn Disease; Margins of Excision; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellvizio (Experimental): Cellvizio is a confocal laser endomicroscopy providing the possibility of obtaining in vivo high-magnification images of the gut epithelium. This allows real-time examination of the gastrointestinal mucosa at the cellular and subcellular level
  Interventions: Procedure: cellvizio

INTERVENTIONS:
Procedure: cellvizio — During surgery an intravenous injection of fluorescein will be performed. The surgeon will, then, evaluate the ileal section margins on the mucosa, the serosa and the mesentery to evaluate if the section margin in microscopically inflammatory or not. She/he will then evaluate (in cm) the length between this section margin and the theorical section margin to be on a non-inflammatory tissue on the mucosa, serosa and mesentery. The data will be filled during surgery, blind from the pathological analysis. The pathological analysis will also be blind from the Cellvizio data. A video collection will be performed anonymously.

SUMMARY:
Crohn disease is an inflammatory bowel disease. A surgical procedure is required in about 80% of cases. Surgery doesn't cure from Crohn's disease but the type of surgery remains important as there are several intraoperative risk factors for recurrence. Among these factors the microscopic inflammation at the resection margins. This is a crucial point, if the resection is too large there is a risk of short bowel syndrome, if the resection is too short (microscopic inflammation at resection site), there is a higher risk of postoperative recurrence (75% vs 46% at 18 months). Surgeons have to do a limited resection (2cm from macroscopic crohn disease). However this macroscopic non inflammatory resection margin can be microscopically inflammatory (up to 80%). Thus it is useful to evaluate if there is a microscopic inflammation at the resection margin. Moreover there is an increase interest for the role of the mesentery for recurrence but its role remains unclear. It is of interest to clarify the border between the inflammatory and non-inflammatory mesentery. Cellvizio is a confocal laser endomicroscopy providing the possibility of obtaining in vivo high-magnification images of the gut epithelium. This allows real-time examination of the gastrointestinal mucosa at the cellular and subcellular level. Cellvizio has never been used during surgery for Crohn disease.

The aim of this study is to evaluate the intraoperative use of Cellvizio (using the CelioFlex microsonde) with an intravenous injection of fluorescein to determine the best ileal resection margins in Crohn disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need a ileocaecal resection for a Crohn disease whatever is the phenotype of the Crohn's disease

Exclusion Criteria:

* Patients<18 years old,
* pregnancy or breastfeeding,
* patients who have an ileocolic resection for a surgical recurrence of the Crohn's disease.
* Patients operated in emergency for a peritonitis,
* patients who have a contra-indication for fluorescein injection or severe allergia to any drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
concordance between the Cellvizio pictures and the pathology incidence | 2 years
  concordance between the Cellvizio pictures and the pathology for microscopic inflammation at the ileal resection margin.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No